CLINICAL TRIAL: NCT01923194
Title: A Randomized, Assessor-blinded, Parallel Group, Multi-center, Non-inferiority Study Investigating the Efficacy and Safety of Highly Purified Urofollitropin for Injection Compared to Recombinant Human Follitropin Alfa for Injection for Ovulation Induction Using a Low-dose, Step-up Protocol in Chinese Females With WHO Group II Anovulatory Infertility Failing to Conceive on Clomiphene Citrate
Brief Title: Evaluation of Efficacy and Safety of Highly Purified Urofollitropin for Ovulation Induction in Chinese Females
Acronym: Compass
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000055
Record Dates: First submitted 2013-08-12; First posted 2013-08-15 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Anovulation
MeSH Terms: conditions — Anovulation | interventions — Urofollitropin; follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Drug: Highly Purified Urofollitropin
- Comparator Group (Active Comparator)
  Interventions: Drug: Recombinant Human Follitropin Alfa

INTERVENTIONS:
Drug: Highly Purified Urofollitropin — for Injection
  Other Names: Bravelle®
  Arms: Test Group
Drug: Recombinant Human Follitropin Alfa — for Injection
  Other Names: Gonal-F®
  Arms: Comparator Group

SUMMARY:
Evaluate the Efficacy and Safety of Highly Purified Urofollitropin for Injection Compared to Recombinant Human Follitropin Alfa for Injection for Ovulation Induction in Chinese females

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form prior to screening evaluations
* Chinese females between the ages of 20-39 years
* Infertility for at least 1 year before screening
* Women WHO type II anovulatory infertility with chronic anovulation (defined as amenorrhoea (i.e., no menstrual bleeding for 6 months or more) or oligoamenorrhoea (i.e., cycles of more than 35 days) ) with progestogen induced withdrawal bleeding or spontaneous menstrual bleeding
* Failure to conceive after at least one cycle of ovulation induction with clomiphene citrate
* Bilateral tubal patency documented by a hysterosalpingography or sonohysterography or laparoscopy within 2 years prior to screening
* Normal pelvis documented by a transvaginal ultrasound with respect to uterus, Fallopian tubes and ovaries within 3 months prior to screening
* Early follicular phase serum levels of FSH within normal limits (1-12 IU/L,) (results obtained within 2 months prior to randomization)
* LH (Luteinizing hormone), prolactin , E2 (estradiol), progesteron, total testosterone, and TSH (thyrotropin) levels within normal limits for the clinical laboratory
* Male partner with a semen analysis obtained within 12 months prior to randomisation and showing acceptable values for semen according to the local laboratory, or showing more than 2.000.000 progressive motile sperm per mL after capacitation (in case of IUI (intrauterine insemination))
* BMI (Body mass index) is ≥ 18.5 and < 30 kg/m2

Exclusion Criteria:

* Any known clinically significant systemic disease
* Known past or current thrombophlebitis or thromboembolism including venous thrombosis disease and active or recent arterial thrombosis disease
* Any known endocrine or metabolic abnormalities which can compromise participation in the trial with the exception of controlled thyroid function disease
* Any known concomitant medications that would interfere with evaluation of study medications. Specifically, any non-study hormonal therapy (except for thyroid medication), anti-psychotics, anxiolytics, hypnotics and sedatives, and need for continuous use of prostaglandin inhibitors (non-steroid anti- inflammatory drugs (NSAIDs), including aspirin) at the time of study entry.
* Known history of 12 or more unsuccessful (no pregnancy achieved) ovulation induction cycles
* Any known treatment with clomiphene citrate, metformin, gonadotropins or GnRH analogues within one month prior to randomisation
* Ovarian cysts with a mean diameter ≥ 15 mm that have persisted for more than one cycle or ovarian endometrioma on ultrasound
* Known at least one previous cycle experienced luteinized unruptured follicle syndrome
* Known abnormal results of cervical examination of clinical significance obtained within 1 years prior to screening
* Abnormal vaginal bleeding of undetermined origin
* Known tumors of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus
* Known malformations of the sexual organs incompatible with pregnancy
* Known current or past (last 12 months) abuse of alcohol or drugs
* Known history of chemotherapy (except for gestational conditions) or radiotherapy
* Finding of any clinically relevant abnormal laboratory value
* Use of any non registered investigational drugs during 3 months before screening or previous participation in the study
* Pregnancy, lactation or contraindication to pregnancy

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The ovulation rate defined as the percentage of subjects who present ovulation | From 6 days up to 7 weeks post hCG (human chorionic gonadotropin) administration

SECONDARY OUTCOMES:
The positive serum progesterone rate | 6~9 days post hCG administration
The positive serum β-hCG/hCG rate | 18~22 days post hCG administration
The clinical pregnancy rate | 6~7 weeks post hCG administration
  Regardless of fetal heart beat
The clinical pregnancy rate | 6~7 weeks post hCG administration
  With fetal heart beat
The ongoing pregnancy rate | 11~12 weeks post hCG administration
The follicular development | On the day of hCG administration
Endometrial thickness | On the day of hCG administration
Total FSH (Follicle-stimulating hormone) dose administered | On the day of hCG administration
Number of FSH treatment days | On the day of hCG administration
Frequency and severity of adverse events | Expected maximum of 6 months
Frequency and severity of injection site reactions | Day 1 up to Day 28 of the ovarian stimulation period
Serum estradiol (E2) levels | On the day of hCG administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (12):
- China (12):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Navy General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Tongji Hospital Tongji Medical College of HUST Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - ShengJing Hospital of China Medical University, Shenyang, Liaoning
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality